CLINICAL TRIAL: NCT03001908
Title: A Comparison of Electromyographic(EMG) Activity & Glenohumeral Motion During Posterior Glide Mobilizations in Healthy & Stiff Shoulders
Brief Title: A Comparison of Electromyographic Activity & Glenohumeral Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Responsible Party: Principal Investigator, Brian T Swanson, Assistant Professor, University of New England
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UNE 052316-013
Record Dates: First submitted 2016-12-01; First posted 2016-12-23 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Orthopedic Disorder
Keywords: shoulder; mobilization; electromyography; imaging ultrasound
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- control oscillation (Active Comparator): control subjects with normal shoulders will undergo the glenohumeral mobilization-oscillation
  Interventions: Other: glenohumeral mobilization-oscillation
- control sustained (Active Comparator): control subjects with normal shoulders will undergo the glenohumeral mobilization-sustained
  Interventions: Other: glenohumeral mobilization-sustained
- stiff oscillation (Experimental): subjects with stiff shoulders will undergo the glenohumeral mobilization-oscillation
  Interventions: Other: glenohumeral mobilization-oscillation
- stiff sustained (Experimental): subjects with stiff shoulders will undergo the glenohumeral mobilization-sustained
  Interventions: Other: glenohumeral mobilization-sustained

INTERVENTIONS:
Other: glenohumeral mobilization-oscillation — posterior glide mobilizations oscillated at 1hz, 4 x 30 seconds
  Other Names: musculoskeletal manipulation
  Arms: control oscillation; stiff oscillation
Other: glenohumeral mobilization-sustained — posterior glide mobilization, sustained 4 x 30 seconds
  Other Names: musculoskeletal manipulation
  Arms: control sustained; stiff sustained

SUMMARY:
Pain pressure measurements, fine wire EMG and real time imaging ultrasound will be used to determine the relationships between motion, pain perception, and mobility in the glenohumeral joint. Muscle activity, joint motion, and pain will be measured pre-post randomized interventions to determine the response to various physical therapy techniques.

DETAILED DESCRIPTION:
To achieve the study aims, 88 adults (44 controls, 44 with stiff shoulders) between the ages of 18-65 will be recruited. The investigators will apply a protocol based on current evidence for effectiveness of mobilizations (4 bouts of 30 sec, oscillatory gr III mobilization @1 Hz vs. 4 bouts of 30 seconds, static gr III mobilization), with interventions determined by randomized blocked assignment. Before and after the intervention, the investigators will assess levels of EMG activity of the posterior rotator cuff during a posterior glide, the force required for the mobilization to reach end range stretch, the amount of humeral head translation on the glenoid via US, and pain pressure thresholds (PPT). The data collected will allow investigators to determine the mechanisms involved in range of motion (ROM) changes and hypoalgesia produced by glenohumeral (GH) joint mobilization in both normal and stiff shoulders by evaluating the main and interaction effects of: the type of mobilization (static vs oscillatory), the magnitude of joint translation via imaging ultrasound, the EMG response of the supraspinatus and infraspinatus muscles, and changes in local and central pain processing observed via PPT testing. These data will allow investigators to evaluate whether motion improvements occur due to mechanical factors (stretch of the capsule observed via change in translation), neurophysiologic factors (change in translation associated with reduction in EMG activity), or both. Concurrent measurements of pain processing by the nervous system (local and central mechanisms) will allow evaluation of whether changes in pain processing occur following oscillatory movements, sustained movements, or both. This information will result in improved understanding of the mechanisms of action of joint mobilization, determination of the efficacy of various modes of mobilization to improve joint translation, and determination of the efficacy of various modes of mobilization to decrease pain.

Data analysis:

All data will be analyzed in aggregate form using quantitative statistics. Descriptive statistics will be utilized for demographic data including age, height, weight, gender, handedness, and side of intervention.

Groups will be measured using tests of difference based on group assignments (normal vs stiff shoulder; sustained vs oscillatory mobilization) comparing peak and root mean squared EMG activity, pain pressure thresholds, force of mobilization, and amount of translation measured via US as well as analysis of interaction effects.

All data will be analyzed using an intention to treat model, and any missing data points were replaced using imputation via means of the group.

All outliers, defined as data points beyond the 95th percentile and identified as outliers during analysis in SPSS, will be Winsorized to minimize the effect of potentially spurious outliers via replacement with the highest non-outlier obtained value for the group.

Descriptive statistics including means, ranges and standard deviations will be assessed for each group condition.

Data will be assessed for the required assumptions for parametric testing/ Analysis of variance(ANOVA) including Mauchly's test of sphericity and the Shapiro-Wilk test of normality. Data not meeting the required assumptions will be assessed with the appropriate non-parametric equivalent test.

Aim 1 will investigate the relationships and within and between group differences in rotator cuff activity (EMG) and posterior glide mobility and mobilization force in the glenohumeral joint in individuals with stiff and normal shoulders based on joint mobilization type.

To analyze within subjects main effects, interaction effects, and second order interaction effects of group and mobilization condition on the DV, three-way between-between-within mixed ANOVAs will be used.

IV: shoulder condition stiff vs normal; oscillation vs static posterior glide; time.

X Repeated measure Dependent variables(DV)s: EMG, US translation, force In the presence of significant three way interactions, post hoc testing to determine simple two way interaction effects will be performed using separate two way ANOVAs Univariate testing will be utilized to determine the presence of simple main effects.

Post hoc analysis will utilize pairwise comparisons in the presence of significant main effects. Bonferroni correction will be utilized due to multiple tests, with comparisons within each simple-simple main effect considered a family of comparisons.

To investigate the relationships between rotator cuff activity (EMG) and posterior glide mobility in individuals with stiff and normal shoulders, point bi-serial correlation will be utilized to assess for meaningful relationships between the following variables:

Mobilization condition x change in EMG, US, force Group (stiff vs control) assignment x change in EMG, US, force Aim 2 will investigate the within and between group differences and relationships between changes in PPT and type of mobilization (static, oscillatory) in individuals with stiff and normal shoulders.

Between group differences will be assessed via ind. t-tests, using the dichotomous independent variables (IV) static vs. oscillatory mobilization, and the DV of PPT measures.

Within group differences will be assessed via paired t-tests, using the dichotomous IV static vs. oscillatory mobilization, and the DV of PPT measures.

ELIGIBILITY:
Inclusion Criteria:

* both healthy volunteers, as well as individuals with shoulder stiffness

Exclusion Criteria:

* shoulder surgery within the past 6 months
* history of shoulder fractures
* rheumatoid arthritis
* osteoporosis
* current pregnancy
* active cancer
* blood clotting or connective tissue disorders
* receiving workman's compensation benefits for your shoulder injury
* pending litigation for your shoulder injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
EMG activity of posterior rotator cuff | Immediate post-intervention
  Fine wire EMG used to measure peak and mean activity of supraspinatus, infraspinatus during mobilization

SECONDARY OUTCOMES:
force applied during mobilization | baseline, immediately post intervention (within 3 minutes)
  force sensor used to determine force required to produce glenohumeral translation, compared pre-post intervention
translation of humeral head | baseline, immediately post intervention (within 3 minutes)
  Real time US imaging to determine amount of translation, assess pre-post intervention changes
pain pressure threshold-bilateral deltoid | baseline, immediately post intervention (within 5 minutes)
  pain pressure threshold at deltoid bilaterally; assessed for changes pre-post intervention
pain pressure threshold-bilateral forearm | baseline, immediately post intervention (within 5 minutes)
  pain pressure threshold at medial forearmbilaterally; assessed for changes pre-post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Swanson, PT, DSc, Principal Investigator — University of New England
Locations (1):
- University of New England, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No